CLINICAL TRIAL: NCT01916980
Title: A Phase III, Multicenter, Open-Label Long-Term Trial to Study the Efficacy and Safety of MK-4117 in Japanese Subjects With Eczema/Dermatitis and Dermal Pruritus.
Brief Title: Efficacy and Safety Study of Desloratadine (MK-4117) in Japanese Participants With Eczema/Dermatitis and Dermal Pruritus (MK-4117-202)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4117-202; 132245 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2013-08-02; First posted 2013-08-06 (Estimated); Results first posted 2014-11-19 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2022-02

CONDITIONS: Eczema; Dermatitis; Dermal Pruritus
Keywords: Dermatitis; Dermatitis, Atopic; Skin Diseases; Skin Diseases, Genetic; Genetic Diseases, Inborn; Skin Diseases, Eczematous; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases
MeSH Terms: conditions — Eczema; Dermatitis; Dermatitis, Atopic; Skin Diseases; Skin Diseases, Genetic; Genetic Diseases, Inborn; Skin Diseases, Eczematous; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases | interventions — desloratadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desloratadine: Eczema/Dermatitis (Experimental): Participants with eczema/dermatitis receive desloratadine 5 mg, taken as one 5-mg tablet, orally once daily in the evening for up to 12 weeks. After Week 4, the dose of desloratadine can be increased from 5 mg/day to 10 mg/day (two 5-mg tablets, orally once daily in the evening for up to 8 weeks), if criteria for dose up-titration are met, there is insufficient antipruritic efficacy and there is no safety concern.
  Interventions: Drug: Desloratadine 5 mg
- Desloratadine: Dermal Puritus (Experimental): Participants with dermal pruritus receive desloratadine 5 mg, taken as one 5-mg tablet, orally once daily in the evening for up to 12 weeks. After Week 4, the dose of desloratadine can be increased from 5 mg/day to 10 mg/day (two 5-mg tablets, orally once daily in the evening for up to 8 weeks), if criteria for dose up-titration are met, there is insufficient anti-pruritic efficacy and there is no safety concern.
  Interventions: Drug: Desloratadine 5 mg

INTERVENTIONS:
Drug: Desloratadine 5 mg — Desloratadine 5 mg/day: one 5-mg tablet taken orally once daily in the evening for up to 12 weeks (Desloratadine 10 mg/day: two 5-mg tablets taken orally once daily in the evening for up to 8 weeks)

SUMMARY:
This is an efficacy and safety study of up to 12 weeks of desloratadine in Japanese participants with eczema/dermatitis and dermal pruritus. The primary hypothesis of this study is that the sum of the daytime and nighttime pruritus/itch scores for both the eczema/dermatitis group and the dermal pruritus group will be significantly improved at Week 2 compared to Baseline.

ELIGIBILITY:
Inclusion Criteria:

* Eczema/dermatitis (acute eczema, chronic eczema, contact dermatitis, atopic dermatitis, nummular eczema, seborrheic dermatitis, asteatotic eczema, neurodermatitis, etc. among eczema/dermatitis for which the observation of pruritus is appropriate)
* Dermal pruritus (generalized dermal pruritus, localized dermal pruritus)

Exclusion Criteria:

* Hypersensitivity to antihistamines or ingredients of a study drug

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2013-08-27 (Actual); Primary Completion 2014-03-08 (Actual); Study Completion 2014-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Furue M, Maeda Y, Oshima N, Hisada S. A Phase III clinical trial of desloratadine in Japanese subjects with eczema/dermatitis and cutaneous pruritus: An open label long-term trial. J Clin Therapeut Med. 2016;32(11):877-889.. [in Japanese] https://mol.medicalonline.jp/archive/search?jo=an9cltmd&ye=2016&vo=32&issue=11

RESULTS

PARTICIPANT FLOW:
Groups:
- Desloratadine: Eczema/Dermatitis: Participants with eczema/dermatitis receive desloratadine 5 mg, taken as one 5-mg tablet, orally once daily in the evening for up to 12 weeks. After Week 4, the dose of desloratadine can be increased from 5 mg/day to 10 mg/day (two 5-mg tablets, orally once daily in the evening for up to 8 weeks), if criteria for dose up-titration are met, there is insufficient anti-pruritic efficacy and there is no safety concern.
- Desloratadine: Dermal Pruritus: Participants with dermal pruritus receive desloratadine 5 mg, taken as one 5-mg tablet, orally once daily in the evening for up to 12 weeks. After Week 4, the dose of desloratadine can be increased from 5 mg/day to 10 mg/day (two 5-mg tablets, orally once daily in the evening for up to 8 weeks), if criteria for dose up-titration are met, there is insufficient anti-pruritic efficacy and there is no safety concern.
Period: Overall Study
Arm/Group | Desloratadine: Eczema/Dermatitis | Desloratadine: Dermal Pruritus
Started | 65 | 29
Completed | 58 | 25
Not Completed | 7 | 4
Not completed — Adverse Event | 4 | 2
Not completed — Lack of Efficacy | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Desloratadine: Eczema/Dermatitis | Desloratadine: Dermal Pruritus | Total
Number analyzed (Participants) | 65 | 29 | 94
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.0 (15.2) | 44.1 (21.5) | 36.4 (18.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 17 | 51
  Male | 31 | 12 | 43
Investigator-assessed Sum of Daytime and Nighttime Pruritus/Itch Scores at Baseline [Mean (Standard Deviation); unit: Score on a Scale] — The Investigator assessed the severity of participant pruritus/itch during the daytime (0=Virtually no itching to 4=Cannot relax because of constant itching) and nighttime (0=Virtually no itching to 4=Cannot sleep because of itching) at Baseline. The sum of the daytime and nighttime pruritus/itch scores could range from 0 to 8, with a higher sum score indicating greater severity. Baseline values were assessed based on the participant diary for two days before the Baseline clinic visit and on the participant interview at the Baseline clinic visit.
  Score on a Scale | 4.75 (1.10) | 5.10 (1.47) | 4.86 (1.23)
Participant-assessed Pruritus Visual Analog Scale (VAS) Score at Baseline [Mean (Standard Deviation); unit: Score on a Scale] — Participants assessed the degree of their pruritus using a 100-mm visual analog scale (VAS; 0mm=No itch, 100mm=Worst imaginable itch) at Baseline. Pruritus VAS scores could range from 0 to 100, with a higher score indicating more severe itching. Baseline was defined as the participant evaluation at the day before the Baseline clinic visit.
  Score on a Scale | 60.42 (18.94) | 60.79 (24.45) | 60.53 (20.66)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pruritus/Itch Score (Sum of Daytime and Nighttime Scores) Assessed by the Investigator at Week 2
Description: The Investigator assessed the severity of participant pruritus/itch during the daytime (0=Virtually no itching to 4=Cannot relax because of constant itching) and nighttime (0=Virtually no itching to 4=Cannot sleep because of itching). The sum of the daytime and nighttime pruritus/itch scores could range from 0 to 8, with a higher sum score indicating greater severity. The change from Baseline in the sum of the daytime and nighttime pruritus/itch scores at Week 2 clinic visit was calculated.
Time Frame: Baseline Visit and Week 2 Visit
Population: The Full Analysis Set (FAS) population consisted of all participants who received at least one dose of study drug and had a Baseline or at least one post-Baseline observation for Investigator-assessed pruritus/itch score.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Desloratadine: Eczema/Dermatitis | Desloratadine: Dermal Pruritus
Number analyzed (Participants) | 65 | 29
Score on a Scale | -1.63 [-2.01 to -1.25] | -2.17 [-2.74 to -1.61]
Statistical Analysis 1: Comparison: Desloratadine: Eczema/Dermatitis; Analysis of the change from Baseline in least squares (LS) mean for the Desloratadine: Eczema/Dermatitis group; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis; Model includes terms of visit, group and visit by group interaction; visit is treated as a categorical variable
Statistical Analysis 2: Comparison: Desloratadine: Dermal Pruritus; Analysis of the change from Baseline in LS mean for the Desloratadine: Dermal Pruritus group; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis; Model includes terms of visit, group and visit by group interaction; visit is treated as a categorical variable

2. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event (AE)
Description: An AE is any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug or protocol-specified procedure, whether or not considered related to the study drug or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of the study drug is also an AE.
Time Frame: Up to 14 weeks (Up to 2 weeks after last dose dose of study drug)
Population: The All-Participants-as-Treated (APaT) population consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Desloratadine: Eczema/Dermatitis | Desloratadine: Dermal Pruritus
Number analyzed (Participants) | 65 | 29
Percentage of Participants | 53.8 | 48.3

3. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an AE
Description: as for outcome 2
Time Frame: Up to 12 weeks
Population: The APaT population consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Desloratadine: Eczema/Dermatitis | Desloratadine: Dermal Pruritus
Number analyzed (Participants) | 65 | 29
Percentage of Participants | 6.2 | 6.9

4. Secondary Outcome: Change From Baseline in Pruritus/Itch Score (Sum of Daytime and Nighttime Scores) Assessed by the Investigator at Day 3, Week 1, Week 4, Week 6, Week 8 and Week 12
Description: The Investigator assessed the severity of participant pruritus/itch during the daytime (0=Virtually no itching to 4=Cannot relax because of constant itching) and nighttime (0=Virtually no itching to 4=Cannot sleep because of itching). The sum of the daytime and nighttime pruritus/itch scores could range from 0 to 8, with a higher sum score indicating greater severity. The changes from Baseline in the sum of the daytime and nighttime pruritus/itch scores at the Day 3, Week 1, Week 4, Week 6, Week 8 and Week 12 clinic visits were calculated.
Time Frame: Baseline Visit and Day 3 Visit, Week 1 Visit, Week 4 Visit, Week 6 Visit, Week 8 Visit, Week 12 Visit
Population: The FAS population consisted of all participants who received at least one dose of study drug and had a Baseline or at least one post-Baseline observation for Investigator-assessed pruritus/itch score.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Desloratadine: Eczema/Dermatitis | Desloratadine: Dermal Pruritus
Number analyzed (Participants) | 65 | 29
Score on a Scale
  Change from Baseline at Day 3 (n=65, 29) | -0.83 [-1.18 to -0.49] | -1.59 [-2.10 to -1.07]
  Change from Baseline at Week 1 (n=65, 29) | -1.29 [-1.66 to -0.92] | -2.07 [-2.62 to -1.52]
  Change from Baseline at Week 4 (n=63, 28) | -1.88 [-2.29 to -1.47] | -2.39 [-3.01 to -1.78]
  Change from Baseline at Week 6 (n=62, 26) | -2.33 [-2.72 to -1.94] | -2.48 [-3.07 to -1.89]
  Change from Baseline at Week 8 (n=61, 25) | -2.18 [-2.59 to -1.76] | -3.15 [-3.79 to -2.52]
  Change from Baseline at Week 12 (n=58, 25) | -2.51 [-2.89 to -2.14] | -3.47 [-4.04 to -2.90]

5. Secondary Outcome: Percentage of Participants With Moderate or Remarkable Improvement in the Global Improvement Rate of Pruritus/Itch Assessed by the Investigator at Day 3, Week 1, Week 2, Week 4, Week 6, Week 8 and Week 12
Description: The global improvement judgment criteria were used to assess overall improvement in pruritus/itch. The Investigator assessed the degree of severity of pruritus/itch based on 5 grades (1=Remarkably improved to 5=Aggravated) at Baseline and subsequent clinic visits. The percentages of participants who were remarkably improved (Grade 1=Pruritus/itch disappeared) or moderately improved (Grade 2=Pruritus/itch was greatly improved) at the Day 3, Week 1, Week 2, Week 4, Week 6, Week 8 and Week 12 clinic visits were calculated.
Time Frame: Baseline Visit and Day 3 Visit, Week 1 Visit, Week 2 Visit, Week 4 Visit, Week 6 Visit, Week 8 Visit, Week 12 Visit
Population: The FAS population consisted of all participants who received at least one dose of study drug and had a Baseline or at least one post-Baseline observation for Investigator-assessed Global Improvement.
Measure: Number; unit: Percentage of Participants
Arm/Group | Desloratadine: Eczema/Dermatitis | Desloratadine: Dermal Pruritus
Number analyzed (Participants) | 65 | 29
Percentage of Participants
  Day 3 | 16.9 | 34.5
  Week 1 | 29.2 | 51.7
  Week 2 | 33.8 | 51.7
  Week 4 | 50.8 | 62.1
  Week 6 | 60.0 | 62.1
  Week 8 | 63.1 | 62.1
  Week 12 | 69.2 | 62.1

6. Secondary Outcome: Change From Baseline in the Pruritus/Itch Visual Analog Scale (VAS) Score Recorded by Participants at Day 3, Week 1, Week 2, Week 4, Week 6, Week 8 and Week 12
Description: Participants assessed the degree of their pruritus using a 100-mm visual analog scale (VAS; 0mm=No itch, 100mm=Worst imaginable itch) at Baseline and subsequent clinic visits. Pruritus/itch VAS scores could range from 0 to 100, with a higher score indicating more severe pruritus/itching. The changes from Baseline in the VAS scores for pruritus/itch at the Day 3, Week 1, Week 2, Week 4, Week 6, Week 8 and Week 12 clinic visits were calculated.
Time Frame: Baseline Visit and Day 3 Visit, Week 1 Visit, Week 2 Visit, Week 4 Visit, Week 6 Visit, Week 8 Visit, Week 12 Visit
Population: The FAS population consisted of all participants who received at least one dose of study drug and had a Baseline or at least one post-Baseline observation for participant-assessed pruritus/itch VAS score.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Desloratadine: Eczema/Dermatitis | Desloratadine: Dermal Pruritus
Number analyzed (Participants) | 65 | 29
Score on a Scale
  Change from Baseline at Day 3 (n=65, 29) | -10.03 [-15.22 to -4.84] | -21.90 [-29.66 to -14.13]
  Change from Baseline at Week 1 (n=65, 29) | -12.17 [-17.92 to -6.42] | -24.72 [-33.33 to -16.12]
  Change from Baseline at Week 2 (n=63, 29) | -18.95 [-25.18 to -12.72] | -28.45 [-37.72 to -19.18]
  Change from Baseline at Week 4 (n=63, 28) | -22.36 [-29.01 to -15.71] | -27.74 [-37.66 to -17.82]
  Change from Baseline at Week 6 (n=62, 26) | -27.26 [-33.20 to -21.32] | -30.71 [-39.70 to -21.72]
  Change from Baseline at Week 8 (n=61, 25) | -29.87 [-36.55 to -23.20] | -32.44 [-42.60 to -22.29]
  Change from Baseline at Week 12 (n=58, 25) | -33.02 [-39.65 to -26.39] | -38.74 [-48.76 to -28.73]

ADVERSE EVENTS:
Time Frame: Up to 14 weeks (Up to 2 weeks after last dose of study drug)
Arm/Group | Desloratadine: Eczema/Dermatitis | Desloratadine: Dermal Pruritus
Serious Adverse Events (participants affected / at risk) | 1/65 | 0/29
Other Adverse Events (participants affected / at risk) | 16/65 | 6/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desloratadine: Eczema/Dermatitis (N=65) | Desloratadine: Dermal Pruritus (N=29)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desloratadine: Eczema/Dermatitis (N=65) | Desloratadine: Dermal Pruritus (N=29)
Nasopharyngitis (Infections and infestations) | 13 (16) | 4 (4)
Somnolence (Nervous system disorders) | 4 (4) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.